CLINICAL TRIAL: NCT06335641
Title: Head COOLing in IscHemic Stroke Patients Undergoing EndovAscular Thrombectomy: a Feasibility and Safety StuDy
Acronym: COOLHEAD-2a
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, William Diprose, Clinical fellow, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COOLHD24-CAN / A+10019; ACTRN12621001346864 (Other: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Stroke, Acute
Keywords: Hypothermia; Large vessel occlusion; Neuroprotection
MeSH Terms: conditions — Stroke; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): Head cooling
  Interventions: Device: External active conductive head cooling

INTERVENTIONS:
Device: External active conductive head cooling — Cooling is applied during the endovascular thrombectomy procedure for a maximum of 120 minutes

SUMMARY:
This is an investigator-initiated, prospective, open-label, single-arm, non-randomized study to assess the safety and feasibility of external active conductive head cooling during endovascular thrombectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

- All patients with anterior circulation acute ischemic stroke planned to undergo endovascular thrombectomy will be screened for recruitment.

Exclusion Criteria:

* Admission core body temperature <35°C.
* Known contraindications to hypothermia, including hemodynamically unstable patients, new/symptomatic arrhythmia, hematological dyscrasias that affect thrombosis (cryoglobulinemia, sickle cell disease, serum cold agglutinins), or vasospastic disorders such as Raynaud's or thrombo-angiitis obliterans.
* Skin lesions not allowing secure application of the cooling cap.
* Unable to participate in follow-up at 3 months (e.g., resides outside of Alberta).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
Adherence to the intervention | From time of application in the emergency department until the end of the endovascular thrombectomy procedure
  Adherence is defined as undergoing active conductive head cooling for ≥50% of the time from first application of the cooling device

CONTACTS AND LOCATIONS:
Locations (2):
- Foothills Medical Center, Calgary, Alberta, Canada
- Te Whatu Ora Te Toka Tumai Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided